CLINICAL TRIAL: NCT00216073
Title: A Phase II Trial of Capecitabine, Oxaliplatin and Trastuzumab (CAPOX-T) in Patients With HER-2 Positive Metastatic Breast Cancer: Hoosier Oncology Group BRE03-61
Brief Title: Capecitabine, Oxaliplatin and Trastuzumab in Treating Patients With HER2 Positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patient accrual
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Sanofi (Industry); Hoffmann-La Roche (Industry); Walther Cancer Institute (Other)
Responsible Party: Kathy Miller, M.D., Hoosier Oncology Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG BRE03-61
Record Dates: First submitted 2005-09-09; First posted 2005-09-22 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Oxaliplatin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Capecitabine + Oxaliplatin + trastuzumab. Patients must be HER2 positive.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Trastuzumab

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 825 mg/m2 po bid, days 1-14
Drug: Oxaliplatin — Oxaliplatin 100 mg/m2 IV, day 1
Drug: Trastuzumab — Trastuzumab 6mg/kg IV, day 1. 8 mg/kg loading dose given in cycle 1 for patients without previous trastuzumab therapy only.

SUMMARY:
In vitro data suggest synergy between oxaliplatin and 5-FU. The combination of oxaliplatin with 5-fluorouracil produced objective response rates ranging from 27-34% in two studies of patients with prior chemotherapy. Capecitabine was designed as an orally administered, tumor selective fluoropyrimidine, preferentially converted to 5-FU at the tumor site by the higher levels of pyrimidine nucleoside phosphorylase (PyNPase) in tumor tissues compared to normal tissues. The end result is higher concentrations of 5-fluorouracil in tumor relative to surrounding normal tissue. Trastuzumab is synergistic in vitro with multiple chemotherapeutic agents including the platinum compounds. Studies have shown the efficacy of trastuzumab combined with chemotherapy in patients with HER2 overexpressing metastatic breast cancer. This trial will investigate the activity of capecitabine and oxaliplatin administered with trastuzumab (CAPOX-T) in patients with HER2 overexpressing in patients with advanced disease.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* CAPOX-T (21 day cycle):Capecitabine 825 mg/m2 orally twice daily Days 1-14Oxaliplatin 100 mg/m2 intravenously Day 1
* Trastuzumab : 6 mg/kg intravenously Day 1.8mg/kg loading dose should be given in cycle 1 for patients without previous trastuzumab therapy only.

Patients may continue combination therapy until progression or toxicity intervenes. Patients who discontinue either or both cytotoxic agents due to toxicity may, at the investigators discretion, continue therapy with the remaining agents on study until progressive disease

ECOG performance status 0 or 1

Hematopoietic:·

* ANC > 1,200/mm3·
* Platelets > 100,000/mm3

Hepatic:·

* Total bilirubin < 1.5 x ULN·
* AST < 2 x ULN (up to 5 x ULN in patients with known liver involvement)

Renal:·

* Serum creatinine < 1.5 x ULN and estimated creatinine clearance >50ml/min as calculated with Cockroft-Gault equation

Cardiovascular:·

* No clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.·
* LVEF > LLN by MUGA or ECHO

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of breast cancer with evidence of (1) unresectable, locally recurrent, or (2) metastatic disease.·
* HER2 gene amplification by FISH. HER protein overexpression by immunohistochemistry will not be sufficient for entry.·
* At least one measurable lesion as defined by the RECIST.
* Prior hormonal therapy for metastatic disease is allowed.
* Maximum of one prior chemotherapy regimen or trastuzumab-containing regimen for unresectable, locally recurrent or metastatic disease
* Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.

Exclusion Criteria:

* No prior therapy with capecitabine or oxaliplatin in any setting
* No prior therapy with other platinum compounds·
* No other forms of cancer therapy including radiation, chemotherapy and hormonal therapy within 21 days prior to beginning protocol therapy.·
* No prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil.·
* No prior fluoropyrimidine therapy for metastatic disease is allowed.
* Prior adjuvant fluoropyrimidine therapy is allowed if completed > 12 months from study entry.·
* No symptomatic brain metastasis. ·
* No evidence of serious concomitant systemic disorders incompatible with the study ·
* No peripheral neuropathy ·
* No major surgery within 28 days prior to beginning protocol therapy.·
* Negative pregnancy test·
* No current breastfeeding·
* No malabsorption syndrome·
* No evidence of serious concomitant systemic disorders incompatible with the study·
* Patients must not be treated with any of the following while on protocol therapy or within 28 days prior to beginning protocol therapy: sorivudine, brivudine, cimetidine, allopurinol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-03; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
- · To determine the objective response rate (CR+PR) of capecitabine, oxaliplatin and trastuzumab(CAPOX-T) in patients with HER2 positive metastatic breast cancer. | 18 months

SECONDARY OUTCOMES:
To measure time to progression | 18 months
To determine rate of clinical benefit response (CR + PR + SD > 6 months) | 18 months
To determine toxicity rate of CAPOX-T in this patient population | 18 months
To explore potential correlations between changes in HER2 circulating extracellular domain in the primary tumor with response | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (11):
- United States (11):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - AP&S Clinic, Terre Haute, Indiana
  - Center for Hematology/Oncology of S. Michigan, Jackson, Michigan

REFERENCES:
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/